# Parental stress and disability. A psychological flexibility training programme

ID: CIPI/21/091

Document date: 15<sup>th</sup> November 2021

IP: Francisco Montesinos, Ph.D.

Informed consent form

#### INFORMED CONSENT FORM TO PARTICIPATE IN THE RESEARCH

"Parental stress and disability. A psychological flexibility training programme"

We would like to invite you to participate in this research developed by a team of professors from the Department of Psychology at the European University of Madrid. The programme is aimed at family members (fathers and/or mothers) of legal age who have a child diagnosed with an intellectual disability for more than 6 months, with a good understanding of Spanish, who are not currently or have been in individual and/or group psychological or psychiatric treatment. Participate only if you wish to do so. If you choose not to participate it will not be a disadvantage for you. Before deciding whether you wish to participate, it is important that you understand why this research is being conducted and what your participation involves. Please take the time to read the following information and ask us if anything is unclear or if you would like more information.

#### WHAT DOES THIS STUDY CONSIST OF?

The aim is to evaluate the effectiveness of a psychological intervention programme to see if it helps family members to learn new repertoires to manage general stress levels more effectively, as well as its correlates on physical and psychological health. The results obtained will help us to create effective and efficient intervention protocols for family members in order to offer comprehensive care to the diagnosed child and his/her family unit. They will also help us to see which elements of psychological interventions are useful in order to improve the quality of care. In addition, participation may help you develop a new way of managing stress and coping with the developmental challenges your child faces. At the end of the workshop, you will receive support materials as a guide to what you have learned during the workshop.

## WHAT WILL I BE ASKED TO DO IF I PARTICIPATE IN THIS STUDY?

You will have the possibility to participate in a workshop based on psychological flexibility for three mornings (9 hours in total) in a group format and led by a psychologist-researcher free of charge. You will have to complete some questionnaires before participation, at the end of the programme and 2 months later. Completing the questionnaires will take no more than 15 minutes and will be of immense help to us for the objectives of the study.

## WILL MY INFORMATION BE KEPT PRIVATE?

Your answers will be kept confidential. We will not collect any identifying information. The entire research process will be carried out guaranteeing the anonymity of the participants, and the voluntary nature of participation. The data will be processed in accordance with Royal Decree-Law 5/2018, of 27 July, on urgent measures for the adaptation of Spanish law to European Union regulations on data protection. The data collected will only be accessible to the study researchers. When the results are reported at conferences or in publications, only group summary data will be included, and it will not be possible to identify specific responses.

## WHO CAN I TALK TO IF I HAVE QUESTIONS ABOUT THIS STUDY?

If you need any kind of clarification, you can contact the researchers of this study: David Lobato, at the Department of Psychology of the Universidad Europea, or by email at david.lobato@universidadeuropea.es or by phone at 912115566.

### WHAT ARE MY RIGHTS AS A VOLUNTEER IN A RESEARCH STUDY?

Your participation is completely voluntary. There will be no penalty for you if you choose not to participate. You can stop volunteering at any time you wish.

### WHAT DOES IT MEAN THAT I GIVE MY CONSENT?

That you have understood the information provided on this form and are willing to take part in the study. That you have had a chance to ask the researcher questions and mention any concerns. That the researcher responds to your questions and concerns in an appropriate manner.

Statement of Consent

#### I declare:

1. That I have read and understood all oral and written information regarding participation in the above project. 2. I have had the opportunity to discuss and ask questions about this information and have received appropriate responses from any of the members of the research team conducting this study. 3. I have been assured that the data are confidential. 4. I voluntarily give my consent to participate in this study by attending the workshop for training and completing the questionnaires at the various time points. 5. I give my consent voluntarily and I am aware that I am free to withdraw from the study at any time, for any reason and without explanation.

| l, | | | , with ID |
|---|---|---|---|
| an | d date of birth | consent to my partic | ipation in the study in the terms |
| expressed abo | ove. | | |
| In Madrid on | of | 202 | |